CLINICAL TRIAL: NCT07072039
Title: Evaluation of the Paramedic Evaluation for Acute COPD Exacerbation (PEACE) Intervention
Brief Title: Evaluation of the Paramedic Evaluation for Acute COPD Exacerbation
Acronym: PEACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Laurel O'Connor, Associate Professor of Emergency Medicine, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002240; 1K23HL174454-01A1 (NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Community Paramedicine; Mobile Integrated Health; COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEACE Arm (Experimental): Patients in this arm will receive PEACE Intervention
  Interventions: Procedure: Paramedic Evaluation for acute COPD Exacerbation

INTERVENTIONS:
Procedure: Paramedic Evaluation for acute COPD Exacerbation — The Paramedic Evaluation for Acute COPD Exacerbation (PEACE) program is a mobile integrated health initiative that aims to evaluate and treat COPD exacerbation in the home. The goal of the intervention is to expedite the recognition and treatment of COPD exacerbation as well as For this intervention, ambulatory teams can refer patients for PEACE visits when a patient has been identified as suffering from symptoms consistent with COPD exacerbation. Once a visit is requested via electronic health record order, a community paramedic presents to the patient's home within 2 hours, evaluates the patient using mobile diagnostic testing, and initiates pharmacological therapies protocolized by the pulmonary team. A standardized clinical approach and documentation strategy is used including a focused history and physical exam, venous blood gas, trending pulse-oximetry, and mobile x-ray. The community paramedic is supervised in real-time by an emergency physician to establish a care plan and di

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a serious lung condition that affects millions of people in the United States. Each year, it leads to about 150,000 deaths, nearly 900,000 emergency room visits, and 700,000 hospital stays. When COPD symptoms suddenly get worse-called an exacerbation-it can seriously harm a person's quality of life and often requires emergency care. Treating these flare-ups early can help prevent hospital visits, but right now, there aren't many good ways to make sure people get care quickly.

Mobile Integrated Health (MIH) programs send specially trained paramedics, guided remotely by doctors, to care for patients in their homes. This approach could help people with COPD get faster, more effective care without needing to go to the hospital.

In this project, the investigators are testing a new program called PEACE (Paramedic Evaluation for Acute COPD Exacerbation). The PEACE program sends community paramedics to patients' homes-when needed and in partnership with their regular doctors-to manage worsening COPD symptoms early. The study team will adapt the PEACE program to meet the needs of adults living at home with moderate to severe COPD, gather feedback from patients and healthcare providers, and run a small pilot study to see if the program is practical and helpful.

DETAILED DESCRIPTION:
Evidence-based strategies to ensure that patients with COPD have reliable, timely, equitable access to treatment are lacking. This deficit is particularly evident in communities impacted by determinants of health that adversely impact preventive health behavior and care access.

On-demand Mobile Integrated Health (MIH) teams, comprised of community paramedics supported by centralized physicians, have been developed to care for patients outside of conventional hospital settings. These teams empower physicians to provide enhanced remote care by collecting essential clinical information about patients in their living environment, performing diagnostic testing, and administering therapy in the home. MIH programs decrease emergency medical services utilization and improve patient satisfaction in select populations, but the impact of MIH programs on the outcomes of patients with COPD exacerbation has not been evaluated.

In this project, the study team will implement and refine an MIH intervention for patients living with COPD. The Paramedic Evaluation for Acute COPD Exacerbation (PEACE) intervention will dispatch community paramedics to execute a home-based evaluation and treatment strategy in collaboration with a supervising physician and the patient's ambulatory medical team during and after acute COPD exacerbation to promote wellness and recovery. This intervention is intended to improve clinical outcomes and reduce acute care costs by eliminating barriers to care, generating actionable clinical data that can facilitate appropriate diagnosis, accelerating treatment, and simplifying care coordination. Our central hypothesis, based on preliminary data and input from key informants, is that an intervention that facilitates community-based management of COPD exacerbation will be acceptable and highly adoptable by patients and clinicians.

The Practical Robust Implementation and Sustainability Model (PRISM) implementation framework will be used to describe factors impacting project implementation, with the embedded Expanded RE-AIM (Reach, Effectiveness, Adoption, Implementation, Maintenance) model guiding outcomes measurements. Leveraging our prototypical intervention design, the study team will test and Refine the prototype PEACE intervention in real clinical practice with a cohort of patients who are at high risk of COPD exacerbation. The study team will use a mixed-methods approach to evaluate the usability and acceptability of each operational and clinical component of PEACE. Measures will include a systematic assessment of protocol adherence, survey instruments, and qualitative interviews to explore contextual factors impacting intervention performance. The study team will confirm our findings and adapt the protocols informed by a working group comprised of clinicians and community partners. Up to 25 patient participants will be enrolled in the intervention, plus up to 11 clinician participants will be enrolled to participate in usability/acceptability ratings and qualitative evaluations/focus groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of COPD
2. At least one COPD exacerbation resulting in ED utilization in the six months prior to enrollment
3. COPD GOLD Score letter designation of B, C, or D
4. Receives care in the UMass Memorial Medical Center Pulmonary Clinic or Benedict Family Health Clinic
5. Over 18 years of age
6. Speaks English
7. Resides in the geographical catchment area allowed by the UMass Memorial Medical Center MIH Program's license

Exclusion Criteria:

1. No prior diagnosis of COPD
2. Under 18 years of age
3. Does not speak English
4. Pregnancy
5. Cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | At enrollment
  Ratio of patients enrolled to total patients approached
Reason for Recruitment Refusal | At enrollment
  Reason that approached patients did not enroll in the study
Intervention Acceptability | from enrollment until completion of study activities at 1 year
  Using the healthcare intervention acceptability qualitative framework, investigators will measure intervention acceptability from both patient and clinician perspectives. This validated framework assesses participants' affective attitudes, sense of intervention coherence, self-efficacy, the perceived ethicality of the intervention, intervention burden and anticipated cost, opportunity cost, and perceived effectiveness.
Protocol Fidelity | From enrollment until study completion at 1 year
  Investigators will evaluate adherence to each component of the PEACE protocol by having two independent physician-reviewers audit the EHR and video recordings from every PEACE encounter to ensure that procedures were completed correctly and within the expected timeframe. Particular attention will be focused on visits with operational or clinical "failures," defined as any clinical or operational deviation from intervention protocol or any unexpected ED visit or hospitalization within 72 hours of a PEACE referral.
Sample Retention | From enrollment until completion of study activities at 1 year
  Investigators will track the number of subjects who completed the entire study compared to the number of subjects initially enrolled. The investigators will also evaluate loss to follow-up rate, perceived reason for discontinuation and completeness of post-intervention data collection.
PEACE Referrals | 6 and 12 months after enrollment
  Investigators will track the total number of PEACE referrals requested during the study period

SECONDARY OUTCOMES:
PEACE Disposition | 6 and 12 months after enrollment
  Distribution of participant clinical disposition after PEACE encounter (home versus emergency department)
Unanticipated ED Visits | From enrollment to completion of study activities at 1 year
  ED visits within 72 hours after PEACE visit where patient was treated in place
Hospitalizations | From enrollment until completion of study activities at 1 year
  Number and length of hospitalizations for COPD
Exacerbation Relapse Rate | From enrollment until completion of study activities at 1 year
  Number of occurrences when patients experience worsening COPD symptoms requiring a second pharmacological intervention before resolution of symptoms from a treated exacerbation
COPD-related Medication changes | From enrollment to completion of study activities at 1 year
  Number of adjustments made to study participants' COPD treatment regimen (initiation, discontinuation, dosage adjustment, or substitution of medications aimed at managing COPD)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel O'Connor, MD, MSc, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Clinical and laboratory data: Includes medical history, demographic information, and patient characteristics at enrollment. Other data will be extracted from the electronic health record and patient-facing instruments at 3, 6, and 12 months. This includes healthcare utilization patterns, instances of COPD exacerbation relapse, COPD-related medication adjustments, and mortality. Additionally, patient-reported COPD-related quality-of-life instruments will be captured and tracked throughout the study. These values will be reported as tabular data and stored in a REDCap secure electronic data capture system.
  Interview data: Semi-structured interviews will be performed with patients, clinicians, and administrators. Deidentified, raw transcripts will be generated and coded using methods described in the research strategy. Codebooks will be developed and used for coding transcripts. Codebooks and coding summary files will be shared as detailed below.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Baseline data (data collected before any intervention), such as demographics, that require no additional analyses, will be submitted within 4 months after enrollment is completed. After the study is complete, the study team will submit all remaining scientific data to the data repository and will mark the RCT status as "complete" in clinicaltrials.gov. Under the current repository policies, data will be preserved and available for the wider research community in perpetuity.
Access Criteria: Prior to the release of individual-level data, researchers will be required to complete data sharing and confidentiality agreements as established by the data repository. Researchers must commit to 1) not attempting to re-identify participants, 2) securing the data with appropriate technology and enforcing strict access rules, 3) destroying data after analyses are completed, 4) meeting any requirements as stipulated by the health system involved in the study, and 5) if research is conducted within a covered entity, HIPAA requirements must be met prior to use.

DOCUMENTS (2):
  • Study Protocol (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT07072039/Prot_000.pdf
  • Informed Consent Form (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT07072039/ICF_001.pdf